CLINICAL TRIAL: NCT06235853
Title: Biomarkers of Recurrence and Progression in Non-muscle Invasive Bladder Cancer - an Association With Inflammatory Response and Plasminogen Activation System
Brief Title: Biomarkers of Recurrence and Progression in Non-muscle Invasive Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 0073/DIA/2019/48_KB
Record Dates: First submitted 2024-01-11; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Non-muscle Invasive Bladder Cancer; Cystoscopy; Recurrence; Progression; Bladder Cancer; Biomarkers
Keywords: Non-muscle Invasive Bladder Cancer; Cystoscopy; Recurrence; Progression; Bladder Cancer; Biomarkers
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Recurrence; Disease Progression; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (10 ml) and urine (10 ml) specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients after TURBT with NMIBC: Patients who underwent successful TURBT with histopathological proof of non-muscle invasive bladder cancer. Blood and urine specimen have been gathered prior to hospital admission during visit in out-patient clinic.
  Interventions: Diagnostic Test: Blood serum: sUPAR, PAI-1, IL-8.; Diagnostic Test: Urine: IL-8, APOE, VEGF.

INTERVENTIONS:
Diagnostic Test: Blood serum: sUPAR, PAI-1, IL-8. — The concentration of described biomarkers were measured in serum.
Diagnostic Test: Urine: IL-8, APOE, VEGF. — The concentration of described biomarkers were measured in urine.

SUMMARY:
Bladder cancer (BC) is one of the most common type of cancer globally. Due to its high incidence rate, high risk of recurrence and progression, and frequent cystoscopy surveillance, BC contributes to major healthcare costs across the world. The goal of this prospective study was to evaluate the prognostic value of novel non-muscle invasive bladder cancer (NMIBC) biomarkers for predicting disease recurrence or progression after radical transurethral resection of bladder tumour (TURBT). The data obtained from this study may help physicians identify patients who are at greater risk of NMIBC recurrence or progression and require close supervision.

DETAILED DESCRIPTION:
The aim of our prospective study was to determine the prognostic impact of the inflammatory response and indicators of nutritional status on recurrence and progression of non-muscle invasive bladder cancer (NMIBC) in patients undergoing transurethral resection of bladder tumour (TURBT). We evaluated six biomarkers, 3 in blood serum: soluble urokinase plasminogen activator receptor (sUPAR), plasminogen activator inhibitor-1 (PAI-1), interleukin 8 (IL-8) and 3 in urine: apolipoprotein E (APOE), vascular endothelial growth factor (VEGF), interleukin 8 (IL-8). Furthermore, following indicators of nutritional status were investigated: Glasgow Prognostic Score (GPS) and Modified Glasgow Prognostic Score (mGPS).

The primary endpoint of this study was the recurrence or progression of NMIBC based on the histopathological or cystoscopic result. The study outcome was evaluated during the first surveillance cystoscopy, which was performed in time intervals indicated by European Association of Urology. Based on literature data and statistical assumptions we aimed to recruit 240 patients with NMIBC.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Presence or suspicion of tumour in urinary bladder
* Qualification for the first transurethral resection of bladder tumour

Exclusion Criteria:

1. age < 18 years
2. active urinary tract infection
3. active autoimmune disease
4. end-stage renal failure and renal replacement therapy
5. active hepatitis A, B or C
6. active HIV infection
7. pregnancy
8. factors disqualifying the patient from adjuvant treatment (intravesical immunotherapy or intravesical chemotherapy)
9. bladder tumour stage T2 or more, or urothelial tumour in a location other than the urinary bladder
10. other cancer or systemic anticancer treatment carried out up to 5 years ago
11. factors disqualifying the patient from surgical treatment, e.g. coagulopathies
12. lack of patient consent to collection of blood and urine samples and to follow-up visits

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with suspicion of bladder cancer
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Tumour recurrence or progression | Up to 1 year
  Tumour recurrence or progression based on histopathological result from specimen from follow-up cystoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Klaudia Bardowska, MD, Principal Investigator — Wroclaw Medical University
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be published in open access repository after publication of study results.
Supporting Information: Analytic Code
Time Frame: Unlimited
Access Criteria: Unlimited

REFERENCES:
- [Derived] Bardowska K, Krajewski W, Kolodziej A, Koscielska-Kasprzak K, Bartoszek D, Zabinska M, Chorbinska J, Kubacki F, Krolicki T, Krajewska M, Szydelko T, Kaminska D. Evaluation of six novel biomarkers for predicting recurrence of non-muscle invasive bladder cancer after endoscopic resection- a prospective observational study. World J Urol. 2025 Feb 10;43(1):114. doi: 10.1007/s00345-025-05485-9. PMID 39928162